CLINICAL TRIAL: NCT02179346
Title: Observational Study on the Feasibility, Safety and Efficacy in the Biological Reconstruction of the Hip Joint With Full Thickness Cartilage Defects With an in Situ Polymerizable and Chondrocyte Populated Biomaterial (NOVOCART® Inject)
Brief Title: Observational Study With NOVOCART® Inject in the Reconstruction of the Hip Joint With Full Thickness Cartilage Defects
Acronym: HIP-ACTION
Status: Completed | Type: Observational
Sponsor: Tetec AG (Industry)
Collaborators: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1304
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Cartilage Disease
Keywords: cartilage defect; hip; impingement
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cartilage defects in the hip joint: NOVOCART® Inject Autologous Chondrocyte Implantation

SUMMARY:
Non-interventional study to evaluate safety and efficacy of NOVOCART® Inject in patients with full thickness cartilage defects in the hip.

DETAILED DESCRIPTION:
Prospective and multicenter non-interventional study to evaluate safety and efficacy of NOVOCART® Inject in patients with impingement syndrom in the hip.

Safety: 24-month post treatment follow up period by measuring the number of adverse drug reactions/serious adverse drug reactions.

Efficacy: 24-month post treatment follow up period using iHOT 33 and EuroQuol-5D-5L.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 60 years
* Insulated full thickness cartilage damage of the hip joint after ICRS grade 3
* Received subchondral bone lamella
* received or reconstructed labrum in labrum cartilage defects
* defect size ≥ 1.5 and ≤ 10 cm2
* Intact surrounding cartilage structure around the defect, and the corresponding articular surface
* existence of the written informed consent of the patients after Enlightenment

Exclusion Criteria:

* More than 2 defects or 2 corresponding defects
* defects in both lower extremities simultaneously
* Radiographic signs of osteoarthritis of Kellgren & Lawrence > 1
* Profound bony lesion > 0.5 cm in the defect area
* Presence of rheumatoid, infectious or para-infectious arthritis, as well as state after these diseases
* Skin injury to the limb to be operated on
* cartilage defect of the corresponding articular surface
* Existing medications, drugs or alcohol
* Acute infectious diseases, chronic cardiovascular disease, endocrine or metabolic disorders, autoimmune or neoplastic diseases
* impairment of the upper extremity, which prevents discharge by Crutches
* Known bleeding disorder, such as Hemophilia A / B or thrombophilia
* pregnancy and lactation, which represent the time of treatment is a contraindication
* Known allergy to the ingredients
* inmates in prisons

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: specialist clinical centre
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Number of adverse drug reactions/serious adverse drug reactions as a measurement of safety. | 12 months
  Number of adverse drug reactions/serious adverse drug reactions as a measurement of safety.
Number of adverse drug reactions/serious adverse drug reactions as a measurement of safety. | 24 months
  Number of adverse drug reactions/serious adverse drug reactions as a measurement of safety.

SECONDARY OUTCOMES:
iHOT 33 (international HIP Outcome Tool) as a measurement of function and Quality of life | 12 and 24 months
  Outcome of iHOT 33 as a measurement of function and Quality of life
EQ-5D-5L (5-level EQ-5D ) as a measurement of function and Quality of life | 12 and 24 months
  Outcome of EQ-5D-5L as a measurement of function and Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Klaus-Peter Guenther, Prof. MD, Principal Investigator — Universitätsklinikum Carls Gustav Carus der TU Dresden
Locations (3):
- Germany (3):
  - University Hospital Carl Gustav of TU Dresden, Dresden
  - Essen University Hospital, Essen
  - sporthopaedicum Straubing, Straubing

IPD SHARING:
Plan to Share IPD: No